CLINICAL TRIAL: NCT00003597
Title: A Phase I Study of Thrombopoietin (rhTPO) Plus G-CSF in Children Receiving Ifosfamide, Carboplatin, and Etoposide (I.C.E.) Chemotherapy for Recurrent or Refractory Solid Tumors
Brief Title: Colony-Stimulating Factors in Treating Children With Recurrent or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 09717; CCG-09717; CDR0000066668
Record Dates: First submitted 1999-11-01; First posted 2003-04-18 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Cancer
Keywords: recurrent childhood rhabdomyosarcoma; recurrent renal cell cancer; recurrent neuroblastoma; recurrent childhood liver cancer; recurrent Wilms tumor and other childhood kidney tumors; recurrent retinoblastoma; childhood central nervous system germ cell tumor; recurrent osteosarcoma; recurrent gestational trophoblastic tumor; recurrent malignant testicular germ cell tumor; recurrent intraocular melanoma; recurrent melanoma; unspecified childhood solid tumor, protocol specific; childhood germ cell tumor; recurrent childhood soft tissue sarcoma; recurrent ovarian germ cell tumor; extragonadal germ cell tumor; recurrent uterine sarcoma; neutropenia; thrombocytopenia; recurrent childhood brain stem glioma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood visual pathway glioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood medulloblastoma; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Neoplasms; Carcinoma, Renal Cell; Neuroblastoma; Wilms Tumor; Retinoblastoma; Osteosarcoma; Gestational Trophoblastic Disease; Testicular Neoplasms; Uveal Melanoma; Melanoma; Neutropenia; Thrombocytopenia; Optic Nerve Glioma; Astrocytoma; Medulloblastoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Thrombopoietin; Carboplatin; Etoposide; Ifosfamide; Granulocyte Colony-Stimulating Factor; Filgrastim

ARMS (2):
- Cohort 1 (Experimental): Chemotherapy days 0-4, G-CSF (5 μg/kg/d) as a daily subcutaneous injection beginning on Day 5. All patients receive recombinant human thrombopoietin (rhTPO). rhTPO began on the last day of ICE (Ifosfamide, Carboplatin and Etoposide) chemotherapy (Day 4) and subsequent doses will be administered on Days 6, 8, 10 and 12 (5 doses total). The initial dose of rhTPO was 1.2 μg/kg/dose and was subsequently escalated to 2.4 and 3.6 μg/kg/dose as tolerated. Therapy will continue for maximum six courses. Pharmacokinetic data will be obtained (during course one only).
  Interventions: Biological: recombinant human thrombopoietin; Drug: carboplatin; Drug: etoposide; Drug: ifosfamide; Biological: G-CSF
- Cohort 2 (Experimental): Chemotherapy days 0-4, G-CSF (5 μg/kg/d) as a daily subcutaneous injection beginning on Day 5. All patients receive recombinant human thrombopoietin (rhTPO). The dose of rhTPO 1.2 μg/kg/dose and subsequently escalated to 2.4 and 3.6 μg/kg/dose as tolerated. Patients assigned to Cohort II will receive pre-chemotherapy rhTPO at 3.6 μg/kg/dose on Days -5, -3, -1, and post-chemotherapy rhTPO on Days +4, +6, and +8 (6 doses total. Subsequent courses of chemotherapy will begin as soon as the ANC recovers to
  ≥ 1,000/μL and the platelet count to ≥ 100,000/μL between days 21 and 35. Therapy will continue for maximum six courses. Pharmacokinetic data will be obtained (during course one nly). For the second cohort, full data collection will occur for cycles one and two and limited data collection for cycles 3, 4, 5, and 6.
  Interventions: Biological: recombinant human thrombopoietin; Drug: carboplatin; Drug: etoposide; Drug: ifosfamide; Biological: G-CSF

INTERVENTIONS:
Biological: recombinant human thrombopoietin
  Other Names: RhTPO; BB-IND # 7431)
Drug: carboplatin
  Other Names: Paraplatin; CBDCA; NSC #241240
Drug: etoposide
  Other Names: VP-16; VePesid; NSC #141540
Drug: ifosfamide
  Other Names: IFX; IFOS; NSC #109724; IND #7887
Biological: G-CSF
  Other Names: GRANULOCYTE COLONY-STIMULATING FACTOR; r-metHuG-CSF; Filgrastim; Neupogen®; NSC #614629

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as thrombopoietin and G-CSF may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase I trial to study the effectiveness of colony-stimulating factors in treating children who have recurrent or refractory solid tumors and who are receiving chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the pharmacokinetics and toxicities associated with the administration of recombinant human thrombopoietin in children with solid tumors receiving myelosuppressive chemotherapy with ifosfamide, carboplatin, and etoposide (ICE).
* Determine a safe dose of recombinant human thrombopoietin with filgrastim (G-CSF) in this patient population.
* Evaluate the time to platelet count recovery following chemotherapy in this patient population.
* Evaluate the depth and duration of neutropenia and thrombocytopenia and the number of platelet transfusion events in this patient population.

OUTLINE: This is a dose escalation study of recombinant human thrombopoietin.

All patients receive chemotherapy consisting of carboplatin IV over 60 minutes on days 0 and 1 and etoposide and ifosfamide IV over 60 minutes on days 0-4. Chemotherapy is continued in the absence of disease progression or unacceptable toxicity for a maximum of 6 courses every 21 days.

Cohorts of 3-6 patients each receive escalating doses of recombinant human thrombopoietin IV on days 4, 6, 8, 10, and 12 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which fewer than 2 patients experience dose limiting toxicity. After the MTD is determined an additional cohort of patients are treated at this dose level every other day on days 4-20. Patients receive filgrastim (G-CSF) subcutaneously beginning on day 5 and continuing until absolute neutrophil count is greater than 1000/mm3 for 2 consecutive days or day 33.

PROJECTED ACCRUAL: A total of 24 evaluable patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven (except for brain stem tumors) malignancy that has

failed or relapsed after standard first-line antineoplastic therapy

* Sarcoma (soft tissue and bone)
* Kidney tumors
* Brain tumors
* Other solid tumors (gonadal and germ cell tumors, malignant melanoma,
* retinoblastoma, liver tumors, and miscellaneous tumors) Must have had recurrence within the past 4 weeks

No bone marrow involvement

No prior or concurrent myelogenous leukemia

PATIENT CHARACTERISTICS:

Age:

* 1 to 21

Performance status:

* Lansky or Karnofsky 60-100%

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count greater than 1000/mm3
* Platelet count greater than 100,000/mm3
* No grade III or IV thrombosis

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT less than 2.5 times ULN

Renal:

* Creatinine clearance or glomerular filtration rate at least 70 mL/min

Cardiovascular:

* Ejection fraction normal
* No evidence of arrhythmias requiring therapy
* Fractional shortening greater than 28%

Other:

* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 10 days since prior colony-stimulating factor therapy and recovered
* At least 30 days since prior epoetin alfa
* No other concurrent cytokines, including epoetin alfa

Chemotherapy:

* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas) and
* recovered
* At least 3 months since therapy with etoposide, carboplatin, or ifosfamide
* that is identical to study treatment

Endocrine therapy:

* Not specified

Radiotherapy:

* Concurrent radiotherapy allowed after third course of therapy
* No prior cranial/spinal radiotherapy
* No prior radiotherapy to greater than 50% of bone marrow

Surgery:

* Concurrent surgery allowed after the second course of therapy

Other:

* No concurrent investigational agents
* No concurrent lithium, aspirin, coumadin, or heparin

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 1998-11; Primary Completion 2004-10 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Determine the pharmacokinetics and toxicities associated with the administration of recombinant human thrombopoietin (rhTPO) | length of study
  To determine the pharmacokinetics and toxicities associated with the administration of recombinant human thrombopoietin (rhTPO) in children receiving I.C.E. myelosuppressive chemotherapy.

SECONDARY OUTCOMES:
Evaluate the time for patients to demonstrate platelet recovery | Length of study
  To evaluate the time for patients to demonstrate platelet recovery following I.C.E. chemotherapy with rhTPO + G-CSF.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S. Cairo, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (24):
- United States (23):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital - Kansas City, Kansas City, Missouri
  - Kaplan Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia

REFERENCES:
- [Result] Angiolillo AL, Davenport V, Bonilla MA, van de Ven C, Ayello J, Militano O, Miller LL, Krailo M, Reaman G, Cairo MS; Children's Oncology Group. A phase I clinical, pharmacologic, and biologic study of thrombopoietin and granulocyte colony-stimulating factor in children receiving ifosfamide, carboplatin, and etoposide chemotherapy for recurrent or refractory solid tumors: a Children's Oncology Group experience. Clin Cancer Res. 2005 Apr 1;11(7):2644-50. doi: 10.1158/1078-0432.CCR-04-1959. PMID 15814645
- [Result] Angiolillo A, Krailo M, Davenport V, et al.: A phase I study of thrombopoietin (rhTPO) + G-CSF in children receiving ifosfamide, carboplatin and etoposide (ICE) chemotherapy for recurrent or refractory solid tumors: a Children's Cancer Group (CCG) study. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-1511, 2001.